CLINICAL TRIAL: NCT01639326
Title: Phase II Randomized Pharmacogenetic Study to Evaluate the Efficacy and Safety of FOLFIRI Schedule With High Doses of Irinotecan (FOLFIRI-AD) in Patients With Metastatic Colorectal Cancer According to UGT1A Genotype 1.
Brief Title: Study to Evaluate the Efficacy and Safety of FOLFIRI-AD in Patients With Metastatic Colorectal Cancer UGT1A Genotype 1
Acronym: FOLFIRI-AD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-IRI-2011-134
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2012-06

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Irinotecan high doses (Experimental): Patients will receive irinotecan dose of 300 mg / m² in patients UGT1A1 * 1 / * 1 and 260 mg / m² in patients UGT1A1 * 1 / * 28 intravenous infusion over 90 minutes and folinic acid at a dose of 400 mg / m² intravenous infusion over 2 hours and 5-FU at a dose of 400 mg / m² intravenous bolus and 5-FU 2400 mg / m² intravenous infusion for 46 hours.
  Interventions: Drug: Irinotecan high doses
- Irinotecan standard doses (Active Comparator): Patients will receive irinotecan at a dose of 180 mg / m² intravenous infusion over 90 minutes and folinic acid at a dose of 400 mg / m intravenous infusion over 2 hours and 5-FU at a dose of 400 mg / m² intravenous bolus and 5-FU 2400 mg / m² intravenous infusion for 46 hours
  Interventions: Drug: Irinotecan standard doses

INTERVENTIONS:
Drug: Irinotecan high doses — Irinotecan dose of 300 mg / m² in patients UGT1A1 * 1 / * 1 and 260 mg / m² in patients UGT1A1 * 1 / * 28 intravenous infusion over 90 minutes and folinic acid at a dose of 400 mg / m² intravenous infusion over 2 hours and 5-FU at a dose of 400 mg / m² intravenous bolus and 5-FU 2400 mg / m² intravenous infusion for 46 hours.
  Arms: Irinotecan high doses
Drug: Irinotecan standard doses — Irinotecan at a dose of 180 mg / m² intravenous infusion over 90 minutes and folinic acid at a dose of 400 mg / m intravenous infusion over 2 hours and 5-FU at a dose of 400 mg / m² intravenous bolus and 5-FU 2400 mg / m² intravenous infusion for 46 hours.
  Arms: Irinotecan standard doses

SUMMARY:
This study aims to use the corresponding pharmacogenetic analysis to increase the dose of irinotecan in the schemes commonly used standard chemotherapy in advanced colorectal cancer treatment first. The project aims to improve the therapeutic index of chemotherapy. This optimization is raised based on the administration of different doses of the drug depending on the genotype UGT1A1 gene. The research team proposes this project to demonstrate how the administration of high doses of irinotecan in the FOLFIRI scheme in patients with genotype UGT1A1 favorable (wild homozygous * 1 / * 1 and heterozygous * 1 / * 28), significantly improves the efficiency of the antineoplastic agent without significant increase in toxicity. Secondarily will assess the possible prognostic factors related to tolerance and efficacy.

The primary objective is to evaluate the efficacy of high doses of irinotecan in the FOLFIRI scheme in patients with metastatic colorectal cancer with a favorable genotype UGT1A1 (wild homozygous * 1 / * 1 and heterozygous * 1 / * 28).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic colorectal adenocarcinoma not curable surgically.
* Not received prior systemic therapy for metastatic colorectal cancer. It allows receiving neoadjuvant or adjuvant chemotherapy (without irinotecan) as a treatment of the primary tumor at least six months before inclusion. All toxicities secondary to previous treatment should have been resolved before inclusion. The progression of disease (metastatic disease) should be confirmed radiologically after adjuvant treatment.
* Genotype of the gene UGT1A1 * 1 / * 1 or * 1 / * 28
* Age> or = 18 and <75 years.
* ECOG 0-1.
* Measurable disease according to RECIST version 1.1
* Life expectancy> or equal to 3 months.
* Informed consent, dated and signed.
* Adequate bone marrow function as:

Hemoglobin ≥ 9.0 g / dl (patients with hemoglobin <9 g / dl may be transfused before inclusion in the study) Platelet count ≥ 100 x 109 / L Absolute neutrophil count (ANC) ≥ 1.5x 109 / L - Adequate liver function as: Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN in the absence of liver metastases and ALT and AST ≤ 5 × ULN in the presence of liver metastases Alkaline phosphatase ≤ 2.5 x ULN or ≤ 5 x ULN in the presence of liver metastases or ≤ 10 x ULN in the presence of bone metastases

- Adequate renal function with creatinine levels <1.5 mg / dL. BUN> 50 ml / min

Exclusion Criteria:

* Genotype of the gene UGT1A1 * 28 / * 28 (Gilbert's syndrome)
* Patients who are pregnant or breast-feeding
* Concomitant treatment with other antineoplastic therapy other than specified.
* Patients with active infectious processes and patients with immunosuppressive therapy, or chronic anticoagulant therapy.
* History of malignancy in the last five years except basal cell carcinoma of the skin or carcinoma in situ of the cervix treated properly.
* Patients with positive serology for HIV previously known, chronic diarrhea, inflammatory bowel disease or malabsorption syndrome or tumor obstruction unresolved.
* Clinically significant cardiovascular disease: cerebrovascular accident / stroke (≤ 6 months before inclusion in the trial), myocardial infarction (≤ 6 months before inclusion in the trial), unstable angina, uncontrolled hypertension, congestive heart failure grade II or higher NYHA or serious cardiac arrhythmia.
* Patients with significant neurological or psychiatric disorders, including dementia or poorly controlled epilepsy.
* Patients with any contraindications specified in the Summary of study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2012-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Overall objective response rate (RR) by RECIST criteria v1.1 | 24 months
  The objective response rate, defined as the percentage of subjects who achieved a complete response (CR) or partial (PR) response will be evaluated according to RECIST criteria version 1.1

SECONDARY OUTCOMES:
Adverse Events | 24 months
  The intensity of the adverse reactions are classified according to the system Toxicity Criteria NCI v 4.0.
Progression free survival | 24 months
  Elapsed time from inclusion to the date of documented disease progression or death from any cause (whichever occurs first).
Overall survival | 24 months
  Elapsed time from inclusion to the time when death occurs from any cause. The subjects lost to follow up will be censored at the date of last follow up.
overall response duration | 24 months
  be measured from the date of the first documentation of RP or RC (whatever the state to register first) until the first date to register progression (PG) or death from any cause. Only in this analysis included subjects who achieved a CR or PR.

CONTACTS AND LOCATIONS:
Overall Officials: David Páez, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Montserrat Baiget, MD, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (3):
- Spain (3):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital de Mataró, Mataró, Catalunya/Barcelona
  - Hospital Universitari Mutua de Terrassa, Terrassa, Catalunya/Barcelona